CLINICAL TRIAL: NCT03451019
Title: Effect of Lanthanum Carbonate and Sevelamer Hydrochloride on Gastrointestinal Calcium Absorption in Patients With Moderate to Advanced Chronic Kidney Disease
Brief Title: Different Effects of Non-calcium Phosphate Binders on Serum Calcium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Michal Nowicki, Prof, Medical University of Lodz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S-L2018
Record Dates: First submitted 2018-02-20; First posted 2018-03-01 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease - mineral bone disorder, phosphate-binders
MeSH Terms: conditions — Renal Insufficiency, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Sevelamer; lanthanum carbonate

STUDY DESIGN:
Intervention Model Description: Prospective randomized open-label study included 34 patients with CKD. Single oral dose of one of phosphate binders (sevelamer or lanthanum) were administered in random order 15 minutes after 5 g calcium carbonate with standardized meal. Serum calcium, phosphate and parathormone were measured at 0, 3, 6, 12, 24 hours after each medication. Bone alkaline phosphatase (BAP), sclerostin, calcitriol and FGF-23 were measured at 0, 12 and 24 hours after dose. Calcium and phosphate were measured in 24h urine collections after each drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sevelamer hydrochloride (Active Comparator): the subject receive a single dose of 2,4 g
  Interventions: Drug: Sevelamer Hydrochloride; Drug: Lanthanum Carbonate
- lanthanum carbonate (Active Comparator): the subject receive a single dose of 1.0 g
  Interventions: Drug: Sevelamer Hydrochloride; Drug: Lanthanum Carbonate

INTERVENTIONS:
Drug: Sevelamer Hydrochloride — Single oral doses of lanthanum (1000 mg) or Sevelamer (2400 mg) were administered in random order 15 minutes after 5 g calcium carbonate with standardized meal
  Other Names: Renagel
Drug: Lanthanum Carbonate — Single oral doses of lanthanum (1000 mg)
  Other Names: Fosrenol

SUMMARY:
Sevelamer hydrochloride (SE) can increase intestinal calcium absorption in contrast to lanthanum carbonate (LA). Study compared effect of LA and SE on serum and urine phosphate and calcium, and hormones regulating mineral-bone metabolism.

DETAILED DESCRIPTION:
Recent experimental studies have shown that a non-calcium based phosphate binder sevelamer hydrochloride can increase intestinal calcium absorption in contrast to lanthanum carbonate. It is unknown whether such the difference may have an effect on bone metabolism and/or modify the development of vascular calcification in patients with chronic kidney disease. The aim of the study was to compare the effect of a single dose of 1000 mg of lanthanum carbonate with 2,4 mg of sevelamer hydrochloride on serum and urine calcium following an oral load of 5 g of calcium carbonate given with a meal with standardized phosphate content.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* with eGFR ≤45 ml/min

Exclusion Criteria:

* hypercalcemia (>ULN),
* serum phosphate >1.2 times normal value
* calcium-phosphate disturbances not associated with CKD, e.g. Paget disease, osteoporosis, any bone fracture within 6 months before study, multiple myeloma or any neoplastic disease, liver or biliary tract disease, primary hyperparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
the change of serum calcium for 24 hours after each drug | 3, 6, 12 and 24 hours after administration of each drug
  absolute change vs baseline and 24h area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Michal Nowicki, Prof.MD PhD, Principal Investigator — Medical University of Lodz
Locations (1):
- Department of Nephrology, Hypertension and Kidney Transplantation, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Makowka A, Nowicki M. Different Effect of Lanthanum Carbonate and Sevelamer Hydrochloride on Calcium Balance in Patients with Moderate to Advanced Chronic Kidney Disease. Ther Clin Risk Manag. 2021 Nov 2;17:1145-1151. doi: 10.2147/TCRM.S330649. eCollection 2021. PMID 34754193